CLINICAL TRIAL: NCT07322016
Title: A Single-dose, Open-label Phase I Clinical Trial Comparing the Pharmacokinetics, Safety and Pharmacodynamics of HRS-1301 Tablets in Subjects With Mild, Moderate and Severe Renal Insufficiency and Healthy Subjects
Brief Title: A Study of HRS-1301 Tablets in Healthy Subjects and Those With Impaired Kidney Function
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-1301-103
Record Dates: First submitted 2025-12-19; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Intervention Model Description: The Pharmacokinetics (PK), safety and Pharmacodynamics (PD) characteristics of a single oral administration of HRS-1301 tablets in subjects with mild, moderate and severe renal insufficiency and healthy subjects were compared using a single-dose, open-label design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-1301 Tablet Group (Experimental): Treatment for oral medication.
  Interventions: Drug: HRS-1301 Tablet

INTERVENTIONS:
Drug: HRS-1301 Tablet — HRS-1301 tablet, oral medication.

SUMMARY:
The primary objective of this study is to evaluate pharmacokinetics of HRS-1301 tablets in subjects with impaired kidney function in comparison with healthy subjects, to develop dose recommendations for patients with renal impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the content, process, and possible adverse reactions of the trial;
2. Male or female subjects aged 18 to 65 (including 18 and 65);
3. Body mass index (BMI) ranges from 18 kg/m2 to 30 kg/m2 (including 18 and 30),and Male weight ≥ 50.0 kg, female weight ≥ 45.0 kg;
4. The glomerular filtration rate should meet the following criteria (GFR, mL/min): Subjects with mild renal impairment: 60-89 mL/min; Subjects with moderate renal impairment: 30-59 mL/min; Subjects with severe renal function impairment: 15~29 mL/min.

Exclusion Criteria:

1. Individuals with a specific history of allergies (such as asthma, urticaria, eczema, etc.), or those with an allergic constitution (such as those allergic to any drug or food), or those known to be allergic to any component of the studied drug;
2. Those with cardiogenic shock, severe conduction obstruction, sick sinus syndrome, heart failure (NYHA grade III-IV), persistent rapid arrhythmia, tortuous ventricular tachycardia or ventricular tachycardia at the pointed point, a history of clinically significant T-wave changes, myocardial infarction, or angina pectoris;
3. Suffering from malignant tumors, or having a history of malignant tumors within 5 years prior to screening (excluding skin non-melanomas that have been treated without recurrence signs and resected cervical intraepithelial neoplasia);
4. Those with a history of gastric or intestinal surgery that some researchers believe may affect drug absorption;
5. Those who have suffered severe trauma or undergone major surgical operations within the three months prior to screening, or who plan to undergo surgery during the trial period;
6. Those who have participated in any clinical trials of drugs or medical devices within three months prior to screening, or those who are still within five half-lives of the drug before screening (whichever is longer);
7. Those who have donated blood of ≥ 400 mL within 4 weeks before screening, or have suffered severe blood loss (blood loss ≥ 400 mL), or have received blood transfusion within 8 weeks;
8. Those who received live (attenuated) vaccines within 4 weeks prior to screening or those who plan to receive them during the trial;
9. Those with potential difficulties in blood collection and a history of fainting at the sight of needles or blood;
10. For patients with renal insufficiency,those who have received renal replacement therapy (such as peritoneal dialysis, hemodialysis, etc.) within 3 months prior to the screening or during the expected trial period；
11. For patients with renal insufficiency，screening individuals with underlying diseases that induce chronic kidney disease within the previous three months and are judged by researchers to be poorly controlled, such as diabetic patients with HbA1c > 10%, and hypertensive patients with systolic blood pressure > 180 mmHg and diastolic blood pressure > 120 mmHg, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Maximum concentration (Cmax). | 0 hour to 8 days after dosing.
  Pharmacokinetic parameters of HRS-1301 in plasma.
Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (AUC0-last). | 0 hour to 8 days after dosing.
  Pharmacokinetic parameters of HRS-1301 in plasma.
Area under the concentration-time curve from time zero to infinity (AUC0-inf). | 0 hour to 8 days after dosing.
  Pharmacokinetic parameters of HRS-1301 in plasma.

SECONDARY OUTCOMES:
Time of maximum concentration (Tmax). | 0 hour to 8 days after dosing.
  Pharmacokinetic parameters of HRS-1301 in plasma.
Area under the concentration-time curve from time zero to the end of the dosing interval tau (AUC0-tau). | 0 hour to 8 days after dosing.
  Pharmacokinetic parameters of HRS-1301 in plasma.
Elimination half-life (t1/2). | 0 hour to 8 days after dosing.
  Pharmacokinetic parameters of HRS-1301 in plasma.
Apparent clearance (CL/F). | 0 hour to 8 days after dosing.
  Pharmacokinetic parameters of HRS-1301 in plasma.
Apparent volume of distribution (Vz/F). | 0 hour to 8 days after dosing.
  Pharmacokinetic parameters of HRS-1301 in plasma.
Cumulative drug excretion in urine (Ae,urine). | 0 hour to 6 days after dosing.
  Pharmacokinetic parameters of HRS-1301 in urine.
Cumulative drug excretion fraction in urine (fe,urine). | 0 hour to 6 days after dosing.
  Pharmacokinetic parameters of HRS-1301 in urine.
Incidence of adverse events (AEs). | 0 hour to 8 days after dosing.
  Safety and tolerability.
Incidence of serious adverse events (SAEs). | 0 hour to 8 days after dosing.
  Safety and tolerability.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided